CLINICAL TRIAL: NCT03279302
Title: A Phase 1, Open-Label, Partially Randomized, 3-Part, Parallel Group Trial to Evaluate the Pharmacokinetic Profile of Glepaglutide (ZP1848) After a Single Intravenous Injection and After Multiple Subcutaneous Injections in Healthy Subjects
Brief Title: Trial to Evaluate the PK Profile of Glepaglutide (ZP1848) After a Single IV and After Multiple SC Injections in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZP1848-16182
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A (Experimental): 1 mg glepaglutide once daily, given as single SC injections on Days 1 to 7
  Interventions: Drug: Glepaglutide
- Group B (Experimental): 5 mg glepaglutide once daily, given as single SC injections on Days 1 to 7
  Interventions: Drug: Glepaglutide
- Group C (Experimental): 5 mg glepaglutide once weekly, given as single SC injections on Days 1, 8, 15, 22, 29, and 36
  Interventions: Drug: Glepaglutide
- Group D (Experimental): 10 mg glepaglutide once weekly, given as single SC injections on Days 1, 8, 15, 22, 29, and 36
  Interventions: Drug: Glepaglutide
- Group E (Experimental): 1 mg glepaglutide, given as an IV infusion at a rate of 4 mg/h for 15 minutes on Day 1
  Interventions: Drug: Glepaglutide

INTERVENTIONS:
Drug: Glepaglutide — Solution for injection
  Other Names: ZP1848

SUMMARY:
The primary objective of the trial is to characterize the pharmacokinetic (PK) profiles of glepaglutide and its primary active metabolites following once-daily and once-weekly subcutaneous (SC) injections and after a single intravenous (IV) infusion in healthy subjects.

Glepaglutide is a proposed International Nonproprietary Name for ZP1848

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations
* Body Mass index between 18 and 30.0 kg/m2
* Able to comply with all the trial procedures
* females will not be pregnant or lactating
* If female of childbearing potential or male agree to use contraception as defined in the protocol
* Male subjects must also be willing to refrain from donating sperm from trial Check-in until 90 days after the last dose

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of bowel obstruction, stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and/or cholecystectomy or hernia repair will be allowed).
* Clinically significant abnormality on 12-lead ECG
* Clinically significant abnormality in hematology, clinical chemistry, or urinalysis
* History of alcoholism or drug/chemical abuse within 2 years
* Alcohol consumption of > 21 units per week for males and > 14 units for females
* Positive urine drug screen
* Positive hepatitis panel and/or positive human immunodeficiency test
* Receipt of any investigational product within 30 days or 5 half-lives
* Previous exposure to GLP-1, GLP-2, human growth hormone, or analogs thereof 30 days prior to Check-in
* Use or intend to use any medications/products known to be strong inhibitors or strong inducers of cytochrome P450 3A enzyme, including St. John's wort
* Use of tobacco, smoking cessation products, or products containing nicotine (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine lozenges, or nicotine gum ) within 3 months prior to Screening
* Receipt of blood products within 2 months prior to Check-in and throughout the trial.
* Donation of blood or significant blood loss from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening and throughout the trial.
* Poor peripheral venous access.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter - half life | Day 0 up to Day 73
  Half life of glepaglutide and active metabolites
Pharmacokinetic parameter - total body clearance | Day 0 to Day 22
  Total body clearance after IV administration
Pharmacokinetic parameter - Apparent clearance | Day 0 to Day 73
  CL/F for subcutaneous doses
Pharmacokinetic parameter - Volume of distribution | Day 0- Day 22
  Volume of distribution after IV dosing
Pharmacokinetic parameter - apparent volume of distribution | Day 0 to Day 73
  Vss/F and Vz/F for subcutaneous doses

SECONDARY OUTCOMES:
Pharmacokinetic parameter - Cmax | Day 0 to Day 73
  Maximum observed plasma concentration
Pharmacokinetic parameter - tmax | Day 0 to Day 73
  time of maximum observed plasma concentration
Pharmacokinetic parameter - AUC | Day 0 to Day 73
  Area under the curve
Pharmacodynamic parameter - plasma citrulline levels | Day 0 to Day 73
  change in plasma citrulline levels
ADA incidence | Day 0 to Day 73
  Overall incidence of anti-glepaglutide antibodies
Safety and tolerability - AEs | Day 0 to Day 73
  Incidence, nature, and severity of adverse events, abnormal clinical laboratory tests, and injection site reactions
Safety and tolerability - ECGs | Day 0 to Day 73
  12 lead electrocardiogram parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Covance CRU, Dallas, Texas, United States

REFERENCES:
- [Derived] Agersnap MA, Sonne K, Knudsen KM, Knudsen CB, Berner-Hansen M. Pharmacokinetics of Glepaglutide, A Long-Acting Glucagon-Like Peptide-2 Analogue: A Study in Healthy Subjects. Clin Drug Investig. 2022 Dec;42(12):1093-1100. doi: 10.1007/s40261-022-01210-1. Epub 2022 Nov 2. PMID 36323988